CLINICAL TRIAL: NCT02283320
Title: An Open Label, Multicenter, Phase 2 Study to Determine the Safety and Efficacy of BIND-014 (Docetaxel Nanoparticles for Injectable Suspension) as a Second-Line Therapy for Patients With KRAS Mutation Positive or Squamous Cell Non-Small Cell Lung Cancer
Brief Title: A Study of BIND-014 (Docetaxel Nanoparticles for Injectable Suspension) as Second-line Therapy for Patients With KRAS Positive or Squamous Cell Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BIND Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIND-014-007
Record Dates: First submitted 2014-10-21; First posted 2014-11-05 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: KRAS Positive Patients With Non-small Cell Lung Cancer; Squamous Cell Non-small Cell Lung Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BIND-014 (Docetaxel Nanoparticles for Injectable Suspension) (Experimental)
  Interventions: Drug: BIND-014 (Docetaxel Nanoparticles for Injectable Suspension)

INTERVENTIONS:
Drug: BIND-014 (Docetaxel Nanoparticles for Injectable Suspension)

SUMMARY:
BIND-014 (docetaxel nanoparticles for injectable suspension) is being studied in patients with v-Ki-ras2 Kirsten rat sarcoma viral oncogene homolog (KRAS) mutation positive or squamous cell non-small cell lung cancer (NSCLC) who have progressed after treatment of one prior platinum-containing chemotherapy regimen.

ELIGIBILITY:
Inclusion Criteria:

* Males or females at least 18 years of age
* Diagnosis of NSCLC with locally advanced or metastatic disease
* Positive for KRAS mutation or Squamous cell histology
* Previously treated with one platinum-based chemotherapy
* Disease status must be that of measurable and/or evaluable disease
* Performance status of 0 to 1 on the ECOG Scale
* Prior chemotherapy completed at least 3 weeks prior to study enrollment
* Prior radiation therapy allowed to < 25% of the bone marrow
* Patient compliance and geographic proximity that allow adequate follow-up
* Adequate organ function
* Patients with reproductive potential must use contraceptive methods
* Signed informed consent from patient

Exclusion Criteria:

* Active infection
* Pregnancy or planning to become pregnant
* Breast feeding
* Serious concomitant systemic disorders
* Second primary malignancy
* Patients who are symptomatic from brain metastasis
* Presence of detectable (by physical exam) third-space fluid collections
* More than 1 prior cytotoxic chemotherapy regimen for advanced disease
* Prior treatment with docetaxel
* History of severe hypersensitivity reaction to polysorbate 80
* Peripheral neuropathy at study entry
* Patients known to be HIV positive
* Patients known to be seropositive for hepatitis C hepatitis B
* Congenital long QT syndrome, congestive heart failure, or bradyarrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Disease control rate | Change in tumour size will be assessed using RECIST measurements. RECIST assessments to be carried out at baseline, week 6, week 12 and every 6 weeks thereafter relative to first dose of study drug, an expected average 18 weeks

SECONDARY OUTCOMES:
Progression-free survival | Change in tumor size will be assessed using RECIST measurements. RECIST assessments will be carried out at baseline, week 6, week 12 and every 6 weeks thereafter relative to first dose of study drug, an expected average of 18 weeks.
Overall survival | Participants will be followed for survival, an expected average 24 weeks after treatment discontinuation
Duration of response | Change in tumour size will be assessed using RECIST measurements. RECIST assessments to be carried out at baseline, week 6, week 12 and every 6 weeks thereafter relative to first dose of study drug, an expected average 18 weeks
Time to response | change in tumour size will be assessed using RECIST measurements. RECIST assessments to be carried out at baseline, week 6, week 12 relative to first dose of study drug
Disease control rate | Change in tumour size will be assessed using RECIST measurements. RECIST assessments to be carried out at baseline, week 6, week 12 and every 6 weeks thereafter relative to first dose of study drug, an expected average 18 weeks
Safety and tolerability, as measured by number of participants with adverse events. | Measured from first dose of study drug until 30 days after study discontinuation.
Objective response rate | change in tumour size will be assessed using RECIST measurements. RECIST assessments will be carried out at baseline, week 6, week 12 and every 6 weeks thereafter relative to first dose of study drug, an expected 12 weeks,

CONTACTS AND LOCATIONS:
Locations (32):
- United States (22):
  - Investigative Site: #51, Chandler, Arizona
  - Investigative Site: #30, Goodyear, Arizona
  - Investigative Site: #44, Phoenix, Arizona
  - Investigative Site: #41, Sedona, Arizona
  - Investigative Site: #58, Duarte, California
  - Investigative Site: #47, La Jolla, California
  - Investigative Site: #32, Los Angeles, California
  - Investigative Site: #50, San Francisco, California
  - Investigative Site: #46, Fort Meyers, Florida
  - Investigative Site: #53, Newnan, Georgia
  - Investigative Site: #56, Savannah, Georgia
  - Investigative Site: #35, Zion, Illinois
  - Investigative Site: #36, Las Vegas, Nevada
  - Investigative Site: #60, Portland, Oregon
  - Investigative Site: #34, Pittsburgh, Pennsylvania
  - Investigative Site: # 59, Pittsburgh, Pennsylvania
  - Investigative Site: #39, Amarillo, Texas
  - Investigative Site: #42, Dallas, Texas
  - Investigative Site: 38, Dallas, Texas
  - Investigative Site: #40, Blacksburg, Virginia
  - Investigative Site: #45, Vancouver, Washington
  - Investigative Site: #37, Yakima, Washington
- Russia (10):
  - Investigative Site: #72, Ufa, Bashkortastan
  - Investigative Site: #75, Istra Settle., Moscow Oblast
  - Investigative Site: #74, Arkhangelsk
  - Investigative Site: #78, Kazan'
  - Investigative Site: #70, Moscow
  - Investigative Site: #79, Rostov-on-Don
  - Investigative Site: #76, Saint Petersburg
  - Investigative Site: #71, Saint Petersburg
  - Investigative Site: #73, Saint Petersburg
  - Investigative Site: #77, Saint Petersburg